CLINICAL TRIAL: NCT06589180
Title: Clinical Outcomes of Placenta Previa - an Individualized Scoring System
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Collaborators: Middle-Eastern College of Obstetricians and Gynecologists (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, Chair of Middle-Eastern college of Obstetricians and Gynecologists, senior clinical fellow, principal investigator, Middle-Eastern College of Obstetricians and Gynecologists
Other Study IDs: PPISS
Record Dates: First submitted 2024-08-26; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of the study is to develop a machine learning -based prediction model for patients with placenta previa . The model will be based on patient characteristics, clinical assessment, and disease features to predict disease course, prognosis and establish an individualized plan of care. Individualized management plan comprises timing of delivery, mode of delivery, need for hospital admission, postpartum hemorrhage management plan, and perioperative care.

The primary outcome is to predict maternal complications, primarily major antepartum hemorrhage (APH), defined as blood loss of 50-1000 ml.

DETAILED DESCRIPTION:
• Study settings: This multi-center study will invite at least 8 European-based tertiary centers. Data will be retrospectively collected from January 2018 to December 2023. with a total follow-up of at least 6 weeks postpartum. All women who will be diagnosed with PP during this period will be considered in the study.

• Inclusion Criteria:

* Pregnant women diagnosed with placenta previa at time of routine second trimester ultrasound (18 to 21 weeks of gestation).
* Aged 18 years old or above.
* Diagnosed with PP, followed-up antenatally and delivered within the same center.
* Authorization to use anonymous patient data for research purposes.

Exclusion Criteria:

* Inadequate documentation.
* Non-compliance to antenatal care.
* Previous 1 or more Cesarean deliveries.
* Previous uterine surgeries that approach the uterine cavity (myomectomy).
* Known untreated uterine septum.
* Maternal chronic medical condition that is associated with higher risk of placental insufficiency (including chronic hypertension, pregestational diabetes, chronic renal disease, autoimmune disease).
* Fetal major congenital anomalies.

Data Collection A standardized data collection spreadsheet is designed for this study and will be available for all participating centers. The sheet will comprise drop lists for all nominal, ordinal and binary variables to ensure consistency. Target data will include patient demographics (age, parity, gestational age at diagnosis, mode of conception, body mass index at booking and at delivery, pregnancy interval), hemoglobin at booking, past medical and surgical history, and the presence of any current complications in pregnancy. Diagnostic information including placental location, distance from internal os, the presence of other placental abnormalities as well as diagnostic modality will be collected. Follow-up from the 32-week scan and any subsequent scans will be explored and further follow-up information including hemoglobin levels, bleeding episodes, need for transfusion, administration of steroids, fetal growth, and maternal and neonatal outcomes, will be reviewed, and collected.

Data sheets will be sent on completion to the primary investigators to review and inquire on any unclear entry prior to data cleaning and data analysis.

Secondary outcomes include prediction of need for antenatal transfusion, emergency cesarean delivery, and massive postpartum hemorrhage (defined as blood loss > 2000 ml), and neonatal admission to neonatal intensive care unit (NICU).

ELIGIBILITY:
Inclusion Criteria:

Pregnant women diagnosed with placenta previa at time of routine second trimester ultrasound (18 to 21 weeks of gestation).

Aged 18 years old or above. Diagnosed with PP, followed-up antenatally and delivered within the same center.

Authorization to use anonymous patient data for research purposes

Exclusion Criteria:

Inadequate documentation. Non-compliance to antenatal care. Previous 1 or more Cesarean deliveries. Previous uterine surgeries that approach the uterine cavity (myomectomy). Known untreated uterine septum. Maternal chronic medical condition that is associated with higher risk of placental insufficiency (including chronic hypertension, pregestational diabetes, chronic renal disease, autoimmune disease).

Fetal major congenital anomalies

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Pregnant women diagnosed with placenta previa at time of routine second trimester ultrasound (18 to 21 weeks of gestation).
  Aged 18 years old or above.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-04 (Estimated); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergency cesarean section (CS) | 22 weeks to 37 weeks of gestation
  CS that is indicated earlier than the elective planned date (36-37 weeks of gestation) due to bleeding or preterm labor

SECONDARY OUTCOMES:
Peri-operative blood loss | Time between onset of cesarean section till 24 hours after the procedure
  Amount of blood loss in ml during and up to 24 hours after delivery as measured by suction device and gravimetric measures

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jauniaux E, Alfirevic Z, Bhide AG, Belfort MA, Burton GJ, Collins SL, Dornan S, Jurkovic D, Kayem G, Kingdom J, Silver R, Sentilhes L; Royal College of Obstetricians and Gynaecologists. Placenta Praevia and Placenta Accreta: Diagnosis and Management: Green-top Guideline No. 27a. BJOG. 2019 Jan;126(1):e1-e48. doi: 10.1111/1471-0528.15306. Epub 2018 Sep 27. No abstract available. PMID 30260097
- [Background] Silver RM, Fox KA, Barton JR, Abuhamad AZ, Simhan H, Huls CK, Belfort MA, Wright JD. Center of excellence for placenta accreta. Am J Obstet Gynecol. 2015 May;212(5):561-8. doi: 10.1016/j.ajog.2014.11.018. Epub 2014 Nov 20. PMID 25460838
- [Background] Bowman ZS, Eller AG, Bardsley TR, Greene T, Varner MW, Silver RM. Risk factors for placenta accreta: a large prospective cohort. Am J Perinatol. 2014 Oct;31(9):799-804. doi: 10.1055/s-0033-1361833. Epub 2013 Dec 12. PMID 24338130
- [Background] Ahn KH, Lee EH, Cho GJ, Hong SC, Oh MJ, Kim HJ. Anterior placenta previa in the mid-trimester of pregnancy as a risk factor for neonatal respiratory distress syndrome. PLoS One. 2018 Nov 2;13(11):e0207061. doi: 10.1371/journal.pone.0207061. eCollection 2018. PMID 30388184
- [Background] Silver RM. Abnormal Placentation: Placenta Previa, Vasa Previa, and Placenta Accreta. Obstet Gynecol. 2015 Sep;126(3):654-668. doi: 10.1097/AOG.0000000000001005. PMID 26244528
- [Background] Jing L, Wei G, Mengfan S, Yanyan H. Effect of site of placentation on pregnancy outcomes in patients with placenta previa. PLoS One. 2018 Jul 17;13(7):e0200252. doi: 10.1371/journal.pone.0200252. eCollection 2018. PMID 30016336
- [Background] Feng Y, Li XY, Xiao J, Li W, Liu J, Zeng X, Chen X, Chen KY, Fan L, Chen SH. Relationship between placenta location and resolution of second trimester placenta previa. J Huazhong Univ Sci Technolog Med Sci. 2017 Jun;37(3):390-394. doi: 10.1007/s11596-017-1745-5. Epub 2017 Jun 6. PMID 28585139
- [Background] Sanad AS, Mahran AE, Aboulfotouh ME, Kamel HH, Mohammed HF, Bahaa HA, Elkateeb RR, Abdelazim AG, El-Din MAZ, Shawki HE. The effect of uterine artery ligation in patients with central placenta pevia: a randomized controlled trial. BMC Pregnancy Childbirth. 2018 Aug 29;18(1):351. doi: 10.1186/s12884-018-1989-5. PMID 30157787